CLINICAL TRIAL: NCT01987700
Title: A Randomized, Prospective, Double-blind, Multi-Center Study To Examine And Compare The Outcomes Associated With The Use Of Flex HD®, A Human Acellular Dermal Matrix, And Strattice™, A Porcine Acellular Dermal Matrix Allograft, When Used As A Reinforcing Material In The Repair Of Large Abdominal Wall Hernias By A Component Separation Technique
Brief Title: Multi-Center Study To Examine The Use Of Flex HD® And Strattice In The Repair Of Large Abdominal Wall Hernias
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Musculoskeletal Transplant Foundation (Other)
Collaborators: Washington University School of Medicine (Other); Pines Surgical (Unknown); Meridian Healthcare System (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MTF 01-13
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2015-09

CONDITIONS: Hernia of Abdominal Wall
Keywords: Abdominal Hernia Repair; Dermal Allograft; Mesh; Component Separation
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- FLEX-HD (underlay) (Active Comparator): FLEX-HD human acellular dermal matrix applied using an underlay technique
  Interventions: Device: FLEX-HD
- FLEX-HD (overlay) (Active Comparator): FLEX-HD human acellular dermal matrix applied using an overlay technique
  Interventions: Device: FLEX-HD
- Strattice (underlay) (Active Comparator): Strattice porcine acellular dermal matrix applied using an underlay technique
  Interventions: Device: Strattice
- Strattice (overlay) (Active Comparator): Strattice porcine acellular dermal matrix applied using an overlay technique
  Interventions: Device: Strattice

INTERVENTIONS:
Device: FLEX-HD
  Other Names: Human Acellular Dermal Matrix (HADM)
  Arms: FLEX-HD (overlay); FLEX-HD (underlay)
Device: Strattice
  Other Names: Porcine Acellular Dermal Matrix (PADM)
  Arms: Strattice (overlay); Strattice (underlay)

SUMMARY:
The primary objective of this study is to examine and compare the outcomes associated with the use of Flex HD®, a human acellular dermal matrix (HADM), and Strattice™, a porcine acellular dermal matrix, (PADM) when used as a reinforcing material in the repair of large complicated abdominal wall hernias.

DETAILED DESCRIPTION:
At least 100,000 ventral hernia repairs are performed in the U.S. each year. Recently, biologically-based implants derived from acellular human dermis, porcine small intestinal submucosa, and porcine dermis have been reported in a variety of complex abdominal wall repair procedures. A variety of surgical techniques and implant placement methods have been described, with no one standard technique achieving precedence. Biologic implant reinforcement of a myofascial closure by means of component separation, or at a minimum, where three-layer fascial approximation is not possible, sublay placement (i.e., closure of the posterior rectus sheath under the implant) are described strategies. These techniques allow placement of the implant against an intact fascial layer and may improve implant incorporation into host tissue. However, the current literature shows few, if any, prospective, randomized, head-to-head comparisons of human acellular dermal matrix (HADM) allograft and porcine acellular dermal matrix (PADM) xenograft when used as a reinforcing material in the repair of large abdominal hernias by a component separation technique.

The Musculoskeletal Transplant Foundation (MTF) has manufactured and processed Flex HD Acellular Hydrated Dermis. This acellular dermis is derived from human skin. In complicated ventral hernia repairs, this type of graft tissue is necessary. Flex HD has been shown to reduce operative time, lower operative costs and provides minimal elasticity.

The primary objective of this study is to examine and compare the outcomes associated with the use of Flex HD®, a human acellular dermal matrix (HADM), and Strattice™, a porcine acellular dermal matrix, (PADM) when used as a reinforcing material in the repair of large complicated abdominal wall hernias.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or greater
* Have a BMI <40
* Have a hernia of at least 200 cm^2
* Have no contraindications to test material(s)
* Have a life expectancy greater than 1 year in the opinion of the Investigator
* Able to provide informed consent
* Able and willing to return for scheduled study visits over 1 year post-operatively (following research related surgery)

Exclusion Criteria:

* < 18 years of age
* Subject is determined to have an America Society of Anesthesiologists' (ASA) physical class of 4, 5, or 6.
* Have a BMI > 40
* Have a hernia < 2002 cm
* Have abdominal loss of domain such that the operation would be impractical or would adversely affect respiratory or cardiovascular function to an unacceptable degree in the opinion of the Investigator
* Inability to close the fascia primarily without abdominal wall mobilization or component separation
* Participation in an investigational drug or device study within the past 6 weeks prior to enrollment into this trial
* Have active necrotizing fasciitis or any other known active local or systemic infection
* Have a known collagen metabolism disorder or any medical condition that could interfere with normal tissue healing process as determined by the Investigator
* Have a known active malignancy present and/or had chemotherapy 12 weeks prior to screening or planned chemotherapy within 12 weeks of enrollment with the exception of BCC or SCC
* Have known moderate to severe cirrhosis which in the opinion of the Investigator would impact the outcome of this trial
* Have a life expectancy less than 1 year.
* Be unable to participate in the informed consent process
* Be unable or unwilling to return for scheduled study visits over the 1 year post-operative assessment period
* Subject's ventral hernia is related to an organ transplant surgery
* Received high dose steroids (≥100mg of prednisone) within the past 6 weeks
* Tobacco use within the past 6 weeks or positive serum cotinine test at time of admission
* Uncontrolled diabetes (i.e. known HbA1C value > 7%)
* History of drug addiction (recreational drugs, prescription drugs or alcohol) that in the Investigator's opinion may interfere with protocol assessments and/or the subject's ability to complete the required follow up
* Pregnancy and/or breastfeeding
* Enterocutaneous fistula
* Undergoing concomitant panniculectomy
* Ventral hernia repairs involving actively infected mesh removal
* Inability to obtain primary fascial closure (Intra-operatively)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-25 (Actual)

PRIMARY OUTCOMES:
Incidence of true hernia recurrence (True defect in the mesh/repair in which intra-abdominal contents are protruding through the defect) at or before 1 year | 12 months
  Quantitative data collected over a one-year period:
  * Recurrent hernias requiring surgical intervention
  * Evidence of Eventration/Hernia Recurrence (Radiographic)
  * Fluid collection (Seroma, Hematoma)
  * Surgical Site Infections
  * Systemic Infections
  * Enterocutaneous Fistula
  * Dehiscence
  * Mesh Failure requiring partial or total removal

SECONDARY OUTCOMES:
Incidence of Functional Hernia Recurrence | 12 months
  Subjective comparisons regarding the integrity of repair/eventration/need for reoperation will be based on clinical assessment, photographs, and/ or radiographically.
  1. Eventration ("E") shall be recorded by observing both angles of the photographs taken at expiration and will be classified as: 1) E-Mild: less than 3 cm in both planes, 2) E-Moderate: Between 3 and 5 cm in both planes 3) E- Severe: More than 5cm in both planes.
  2. The need for reoperation ("R") shall be recorded as 1) R-1: Reoperation needed, or 2) R-2: No Reoperation needed. The statistical relationship between these parameters and the repair material (HADM or PADM) will be studied by means of a chi square test.
Patient Satisfaction | 3 months, 6 months, 12 months
  Patient satisfaction ratings via the SF-36 at baseline and at 3, 6, and 12 months following their surgery. Cumulative changes in patient satisfaction will be calculated individually for each patient, collectively for all subjects receiving HADM and for all subjects receiving PADM and then compared collectively to each other.

CONTACTS AND LOCATIONS:
Overall Officials: Grant Bochicchio, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (3):
- United States (3):
  - Pines Surgical, Pembroke Pines, Florida
  - Washington University in St Louis, Barnes Jewish Hospital, St Louis, Missouri
  - CentraState Medical Center, Freehold, New Jersey